CLINICAL TRIAL: NCT03494530
Title: Lixiana Acute Stroke Evaluation Registry
Acronym: LASER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 4.0
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke; Atrial Fibrillation; Hemorrhagic Transformation Stroke
Keywords: atrial fibrillation; ischemic stroke; Hemorrhagic transformation; Edoxaban; cardioembolic stroke; Intracerebral hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Embolic Stroke; Cerebral Hemorrhage | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early initiation of edoxaban (Other): Participants will be initiated on edoxaban within ≤ 5 days following ischemic stroke
  Interventions: Drug: Edoxaban 60 MG; Drug: Edoxaban 30 mg
- Delayed initiation of edoxaban (Other): Participants will be initiated on edoxaban within 6-14 days following ischemic stroke
  Interventions: Drug: Edoxaban 60 MG; Drug: Edoxaban 30 mg

INTERVENTIONS:
Drug: Edoxaban 60 MG — Anticoagulant used to treat atrial fibrillation
  Other Names: Lixiana
Drug: Edoxaban 30 mg — Anticoagulant used to treat atrial fibrillation
  Other Names: Lixiana

SUMMARY:
Study Design:

Lixiana Acute Stroke Evaluation Registry (LASER) is a randomized controlled trial with an associated registry. Patients with previously known or newly diagnosed atrial fibrillation (AF) and acute ischemic stroke within five days will be randomized 2:1 to early (≤ 5 days) or delayed (6-14 days) edoxaban initiation. Ischemic stroke will be defined as evidence of acute focal cerebral infarction confirmed on CT/MRI and/or focal hypoperfusion/vessel occlusion on multimodal CT, or by sudden focal and objective neurological deficits (i.e NIHSS ≥ 1) of presumed ischemic origin persisting > 24 hours.

Study Aim and Objectives:

The primary aim of LASER is to demonstrate the safety of edoxaban initiation within five days of cardioembolic stroke. Secondary aim is to determine predictors of hemorrhagic transformation (HT) after cardioembolic stroke. Investigators will systematically assess prospectively collected Computed Tomography (CT) scan images for evidence of HT and re-infarction.

DETAILED DESCRIPTION:
Study Hypothesis:

Investigators hypothesize that edoxaban initiation within five days of ischemic stroke will not be associated with increased HT rates, relative to patients in whom anticoagulation is delayed. Serial imaging using CT will be utilized to determine the rate of radiological HT after edoxaban initiation. Incident radiological HT rates will be assessed as objective performance criteria for the safety of early versus delayed edoxaban initiation. Investigators also hypothesize that RNA expressed in leukocytes at time of stroke can stratify risk of HT in patients treated with edoxaban. Investigators will assess the rate of recurrent ischemic stroke, but recognize any differences between groups will be hypothesis generating only due to the small trial sample size.

Study Design:

LASER is a randomized controlled, parallel-group, two-arm, assessor-blinded trial with an associated registry. Patients with previously known or newly diagnosed AF-related ischemic stroke within five days will be randomized 2:1 to early (≤ 5 days) or delayed (6-14 days) edoxaban initiation. Ischemic stroke will be defined as evidence of acute focal cerebral infarction confirmed on CT/MRI and/or focal hypoperfusion/vessel occlusion on multimodal CT, or by sudden focal and objective neurological deficits (i.e NIHSS ≥ 1) of presumed ischemic origin persisting > 24 hours. A total of one hundred fifty patients from a comprehensive Canadian stroke center will be enrolled. Eligible patients will be randomized within five days of symptom onset after baseline imaging. Patients with spontaneous parenchymal hemorrhage (PH) (European Cooperative Acute Stroke Study (ECASS) grade PH1 or PH2 on the baseline imaging will not be eligible for randomization. These patients will be included in the registry portion of LASER and follow-up will be identical to that in the trial. The timing of edoxaban initiation in these patients will be at the discretion of the treating physician.

Eligible patients will be randomized 2:1 following open label simple randomization procedure to early (≤ 5 days) or delayed (6-14 days) edoxaban initiation via a centralized web-based randomization process, Research Electronic Data Capture (REDCap, Vanderbilt university). After randomization to early or delayed arms, the decision to time the edoxaban initiation within the specific arm will be at the treating physician's discretion. The rationale for the specific timing of treatment, within the randomization window, will also be recorded by surveying the treating physician in each case.

All randomized patients will be followed for 90 days after edoxaban initiation. A National Institute of Health Stroke Scale (NIHSS) score will be assessed at baseline, 7 and 90 days after edoxaban initiation. Functional outcome will be assessed with a modified Rankin Scale (mRS) score at baseline, 7 and 90 days after edoxaban initiation. Montreal Cognitive Assessment (MoCA) will be performed at baseline, and day 90 after edoxaban initiation. RNA will be used to stratify risk of HT. Functional outcome at 90 days will be dichotomized as favourable (mRS score 0-2) and unfavourable (mRS score 3-6). Quality of life will be assessed with the EuroQol-5 Dimension (EQ-5D) and Visual Analog Scale (VAS) at day 90.

In addition to diagnostic imaging, all patients will have a non-contrast, axial CT scan at baseline (within 24 hours from study recruitment) and at 7±2 days after edoxaban initiation. Therefore, all patients will have a minimum of two scans (diagnostic and pre-randomization).In the event of clinical deterioration, CT scans will be repeated. The original LASER protocol included MRI acquisition in all patients. Following diagnostic CT, all patients were to undergo MRI including diffusion-weighted imaging (DWI to assess the acute infarct volume), Fluid Attenuated Inverse Recovery (FLAIR to assess chronic infarct and white matter ischemic change volumes) and susceptibility weighted imaging (SWI to assess for acute HT and chronic cerebral microbleeds) prior to randomization. Shortly after trial initiation, however, COVID-19 restrictions limited access to research MRI protocols. The protocol was therefore amended and both baseline and day 7 imaging data are limited to CT.

Administrative Structure:

Case report forms and data monitoring will be completed on site. All imaging data will be read centrally at the Stroke Imaging Laboratory at the University of Alberta.

Procedures:

Randomized patients will be treated with edoxaban 60 mg once daily. The edoxaban dose will be reduced to 30 mg once daily if any of the following characteristics are present at the time of randomization or during the study: estimated creatinine clearance (CrCl) of 30 to 50 ml per minute using Cockcroft-Gault Equation or body weight ≤ 60 kg. Prior to edoxaban initiation, all patients will be treated as per the clinical standard of care using antiplatelet(s) and anticoagulation for deep venous thrombosis (DVT) prophylaxis. Any antithrombotic therapy prior to randomization will be recorded.

Imaging Procedures and Analysis:

Anonymized dicom CT data will be assessed by two independent raters, blinded to treatment group, for the presence, number and total volume of regions with infarction. Infarct volumes will be measured using planimetric techniques. Any HT, as well as other intracranial hemorrhage, seen at baseline and day 7 will be graded using the Heidelberg Bleeding Classification (HBC). Incident HT seen on follow-up CT scan is defined as new or progressive HT. Progressive HT will be defined as any increase in the severity grade between the baseline and follow-up scan. Two raters will rate the HT using the Heidelberg criteria.

RNA Analysis:

A blood sample will be drawn into a PAXgene tube for RNA analysis at the time of the baseline CT. RNA will be isolated and measured by RNA sequencing and reverse transcription polymerase chain reaction (RT-PCR). Genes different between patients who develop HT compared to those without HT will be identified by analysis of variance adjusted for covariates as previously described. A prediction model will be developed using the identified genes. The ability of the developed gene model to predict HT will be compared to other factors associated with HT including age, stroke severity, infarct volume.

Endpoints:

The primary study endpoint is the rate of incident (new or progressive) radiological HT. The secondary endpoint is the rate of symptomatic HT, defined as intracerebral hemorrhage within and beyond infarcted brain tissue with PH >1/3 the volume of the ischemic infarct (Class 2 in HBC) associated with clinical deterioration (worsening of NIHSS score by ≥ 4 points) within 30 days of treatment initiation. Other secondary endpoints are recurrent ischemic stroke within 90 days of randomization, recurrent sub-clinical infarcts on follow up CT at 7±2 days post edoxaban initiation, systemic hemorrhagic complication rate within 90 days of randomization, NIHSS at day 7 and 90, mRS score at day 7 and 90, favourable mRS at day 90, and mortality within 90 days, quality of life at 90 days assessed by (EQ-5D) and Visual Analog Scale (VAS), and ability of leukocyte RNA to predict HT.

Investigators will report serious adverse events (SAE) within the study period using standardized event, resolution and association codes, and they will be reported to the local Human Research Ethics Board.

Sample Size:

Based on previous open label studies of DOAC use in acute stroke, the rate of symptomatic HT is likely to be nil, which is why we have made this a secondary endpoint. We have previously demonstrated the rate of asymptomatic HT in serial imaging studies to be as lower as 3% in CT-based studies and up to 13% in MRI based studies. There are no data related to the difference in asymptomatic HT rates in patients randomized to early versus late DOAC initiation. Our aim is to determine the event rates in these two groups with reasonable precision.

A sample size of 150 patients, randomized 2:1 (≤5 days:6-14 days) will allow detection of an asymptomatic hemorrhage rate of 3% (95% CI 0.6-8.5%) in the early treatment arm (n=100) and 4% (95% CI 0.5-13.7%) in the late treatment arm (n=50). Thus, we will have confidence interval width of a maximum of 13.7%, allowing enough precision to demonstrate the safety of early treatment. The rationale for adopting a 2:1 randomization approach is to increase the precision around the estimate of safety in the early treatment arm, without substantively losing power.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients
2. 18 years of age or older
3. Ischemic stroke, diagnosed and enrolled ≤5 days from symptom onset (Ischemic stroke is defined as evidence of acute focal cerebral infarction confirmed on CT/MRI and/or focal hypoperfusion/vessel occlusion on multimodal imaging, or by sudden focal and objective neurological deficits (i.e NIHSS ≥ 1) of presumed ischemic origin persisting > 24 hours)
4. Atrial Fibrillation (AF, paroxysmal or persistent), confirmed with ECG/Holter monitor, or by history (clinical documentation of previous AF must be provided).
5. Informed consent

Exclusion Criteria:

1. Acute or chronic renal failure, defined as eGFR <30 ml/min (Cockcroft Gault formula).
2. Known hypersensitivity to edoxaban.
3. Any significant ongoing systemic bleeding risk, i.e. active GI/GU bleeding or recent major surgery.
4. Recent past history or clinical presentation of ICH, subarachnoid haemorrhage (SAH), arterio-venous malformation (AVM), aneurysm, or cerebral neoplasm.
5. Hereditary or acquired hemorrhagic diathesis.
6. Stroke mimics
7. HT with a grade of parenchymal hemorrhage (PH1 or PH2) on baseline or screening CT. They will be eligible for the registry portion of LASER and follow-up will be identical to that in the trial.
8. Any condition that, in the judgment of the investigator(s), could impose hazards to the patient if study therapy is initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of incident radiological hemorrhagic transformation (HT) | Follow up CT scan at 7±2 days after edoxaban initiation

SECONDARY OUTCOMES:
Rate of symptomatic hemorrhagic transformation (HT) | Within 30 days of edoxaban initiation.
  intracerebral hemorrhage within and beyond infarcted brain tissue with PH >1/3 the volume of the ischemic infarct (Class 2 in HBC) associated with clinical deterioration (worsening of NIHSS score by ≥ 4 points)
Recurrent ischemic events | Within 90 days of randomization
  TIA, ischemic stroke, or systemic emboli
Recurrent sub-clinical infarcts | Follow up CT scan at 7±2 days after edoxaban initiation
  Asymptomatic
systemic hemorrhagic complication rate | Within 90 days of randomization
  Systemic bleeding
NIHSS | At day 7 and 90 after edoxaban initiation
  Clinical assessment of neurological deficits
mRS score | At day 7 and 90 after edoxaban initiation
  Clinical assessment of functional status
favourable mRS at day 90 (mSR 0-2) | At day 7 and 90 after edoxaban initiation
  Clinical assessment of functional status
Mortality | At day 90
  Mortality
EQ-5D and Visual Analog Scale (VAS) | At 90 days after edoxaban initiation
  Quality of life assessment
Ability of leukocyte RNA to predict HT. | Within 3 hours of onset
  Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Brian Buck, MD, Principal Investigator — principle investigator; Ken Butcher, MD, Principal Investigator — Prinicple Investigator
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alrohimi A, Jickling G, Jeerakathil T, Shuaib A, Khan K, Kate M, Hill MD, Buck B, Butcher K. Protocol for LASER: A Randomized Evaluation and an Associated Registry of Early Anticoagulation With Edoxaban After Ischemic Stroke in Patients With Atrial Fibrillation. Front Neurol. 2021 Mar 31;12:645822. doi: 10.3389/fneur.2021.645822. eCollection 2021. PMID 33868150